CLINICAL TRIAL: NCT03801798
Title: A Double-blind, Randomized, Placebo Controlled, Parallel-group, Phase 2a Study to Evaluate the Efficacy and Safety of GC1102 in Combination With Nucleos(t)Ide Analogues (NAs) in Patients With Chronic Hepatitis B
Brief Title: A Study of GC1102(Recombinant Hepatitis B Immunoglobulin) in Chronic Hepatitis B Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Green Cross Corporation (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GC1102B_P2a
Record Dates: First submitted 2019-01-08; First posted 2019-01-14 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Hepatitis B
Keywords: GC1102; GC1102B; Chronic Hepatitis B virus; CHB; NAs; NUC
MeSH Terms: conditions — Hepatitis B; Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NAs antivirals + GC1102 180,000 IU (Experimental): All patients are currently being treated with long-term NA treatment(more than 24 weeks) and will continue using these during the study.
  Each vial contains 1mL of study drug or placebo; Single IV bolus injection of 18mL
  * V2 to V17 : IV bolus injection twice a week
  * V18 to V33 : IV bolus injection once a week
  Interventions: Drug: GC1102
- NAs antivirals + GC1102 Placebo (Placebo Comparator): All patients are currently being treated with long-term NA treatment(more than 24 weeks) and will continue using these during the study.
  Each vial contains 1mL of study drug or placebo; Single IV bolus injection of 18mL
  * V2 to V17: IV bolus injection twice a week
  * V18 to V33: IV bolus injection once a week
  Interventions: Other: GC1102 Placebo

INTERVENTIONS:
Drug: GC1102 — NAs antivirals+GC1102 180,000 IU
  Arms: NAs antivirals + GC1102 180,000 IU
Other: GC1102 Placebo — NAs antivirals+GC1102 Placebo
  Arms: NAs antivirals + GC1102 Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of GC1102 in combination of Nucleo(t)ide analogues (NAs) in patients with chronic hepatitis B

ELIGIBILITY:
Inclusion Criteria:

* Patients who had this study information explained to them and understood it, voluntarily decided participation, and provided written consent
* Patients who Aged ≥19 and ≤ 65 years at the time of signing the consent form
* Patients with chronic hepatitis B who have been taking Nucleos(t)ide analogue antivirals 24 weeks before screening
* Patients whose HBsAg and HBV DNA in blood; 10 IU/mL ≤ HBsAg titer ≤ 1,000 IU/mL and negative(-; below the limit of detection of 10 IU/mL) HBV DNA in the screening test

Exclusion Criteria:

* Patients who have Hepatic diseases (e.g., autoimmune hepatitis) from causes other than hepatitis B
* Patients who have history of liver transplantation, or liver transplantation schedule during the study
* Patients who co-infected with HAV, HCV, HDV and HIV
* Patient with Vasculitis
* Patients who had a loss of blood or donated blood of ≥ 400mL within 8 weeks before the screening
* patient who have active infection(other than chronic hepatitis B infection) requiring continual treatment with antibiotics or antivirals (except for clinically insignificant temporary infection such as cold)

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with ≥ 1log10 reduction in HBsAg titer | from baseline at Week 48 after the first dose of investigational product
  HBsAg titer

SECONDARY OUTCOMES:
Proportions of subjects with ≥ 0.5log10 reduction in HBsAg titer | from baseline at Weeks 12, 24, 36 and 48 after the first dose of investigational product
  HBsAg titer
Proportion of subjects with ≥ 1log10 reduction in HBsAg titer | from baseline at Weeks 12, 24, 36 and 48 after the first dose of investigational product
  HBsAg titer
Change in HBsAg titer | from baseline at Weeks 3, 8, 12, 24, 36 and 48 after the first dose of investigational product
  HBsAg titer
ALT response rates | from baseline at Weeks 12, 24, 36 and 48 after the first dose of investigational product
  Proportions of subjects with ALT ≤ 1.0 X ULN at Weeks 12, 24, 36 and 48 after the first dose of investigational product in subjects with ALT >1.0 X ULN at baseline
HBeAg seroconversion rates | from baseline at Weeks 12, 24, 36 an 48 after the first dose of investigational product
  Proportions of subjects with negative (-) HBeAg result at Weeks 12, 24, 36 and 48 after the first dose of investigational product in subjects with positive (+) HBeAg result at baseline
Rate of HBsAg loss | from baseline at Weeks 12, 24, 28, 36 and 48 after the first dose of investigational product
  Proportions of subjects with negative (-; below the limit of detection of 0.5 IU/mL) HBsAg result at Weeks 24, 28, 36 and 48 after the first dose of investigational product
Proportion of negative (-; below the limit of detection of 10 IU/mL) HBV DNA at each measurement time point | from baseline at Weeks 3, 8, 12, 24, 36 and 48 after the first dose of investigational product
  Proportion of subjects with negative (-; below the limit of detection of 10 IU/mL) HBV DNA at each measurement time point

CONTACTS AND LOCATIONS:
Overall Officials: Sang Hoon Ahn, MD, Principal Investigator — Severance Hospital
Locations (1):
- Severance Hospital, Seoul, South Korea